CLINICAL TRIAL: NCT03791814
Title: A Prospective Cohort Study to Improve HCV Care Using Multidisciplinary Approach to the Treatment of Chronic Hepatitis C in Dialysis Patients: The MATCH-D Study
Brief Title: A Prospective Cohort Study to Improve HCV Care in Dialysis Patients
Acronym: MATCH-D
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped due to difficulty in identifying potential patients.
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Davita Clinical Research (Industry)
Responsible Party: Principal Investigator, Eyob Feyssa, MD, Albert Einstein Healthcare Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MATCH-D study
Record Dates: First submitted 2018-12-31; First posted 2019-01-03 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis C
Keywords: HCV treatment; Zepatier; Dialysis patients
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Zepatier treatment (Experimental): Open-label Zepatier (grazoprevir 100 mg and elbasvir 50 mg) will be administered in this study. Daily treatment of Zepatier for a 12-week duration will be administered.
  Interventions: Drug: Zepatier

INTERVENTIONS:
Drug: Zepatier — Patients screened as HCV positive will receive Zepatier for 12 weeks.

SUMMARY:
Hepatitis C virus (HCV) infects an estimated 185 million individuals worldwide and 3.4 million to 4.4 million people in the United States. Approximately 80% of acutely infected HCV patients progress to chronic infection, 20% of whom develop cirrhosis within 25 years, with 25% of patients with cirrhosis developing hepatocellular carcinoma and/or decompensated liver disease. Hepatitis C virus is the primary cause of liver transplantation in the United States.

There are 6 known genotypes of HCV. The most common genotypes in the United States are genotype 1 (subtypes 1a and 1b), 2, and 3, which together comprise 97% of all infections.

In chronic kidney disease (CKD) patients, the prevalence of HCV infection is higher than in the general population. Patients with impaired kidney function have limited therapeutic options. The US Food and Drug Administration (FDA) recently approved Elbasvir/Grazopevir for treatment of genotype 1 and 4 infection in CKD patients including those on hemodialysis.

At our institution, the Multidisciplinary Approach to the Treatment of Chronic Hepatitis C (MATCH) Initiative is a program which was first implemented to increase screening, diagnosis and treatment of HCV by actively incorporating primary care providers (PCP) at every step of the HCV care process. Following implementation of MATCH, early data indicates, marked increase in screening high risk and baby-boomer cohorts, as well as safe and effective treatment of HCV cases at the primary provider setting. The initiative proved that active participation of PCPs in the care of HCV reduced the treatment lag by 71% compared to traditional care of referring HCV cases to specialized care (Gastroenterology or Hepatology) while keeping similar SVR. We intend to expand the program to improve quality of care for HCV patients in dialysis center. We propose active involvement of dialysis clinical staff including nephrologist, to increase HCV screening rate, promote timely diagnosis and treatment of CHC in patient with end-stage renal disease.

This study is being conducted to evaluate real-world effectiveness of HCV DAA therapy in CHC hemodialysis patients when the DAA-treatment is managed and monitored by the clinical staff of hemodialysis center.

Primary objective: To determine sustained virologic response (SVR) rates attained with open-label Zepatier administered through hemodialysis center under the supervision of a nephrologist in chronic hepatitis C infected (CHC) patient currently on hemodialysis.

Secondary objective:

1. To estimate prevalence of HCV infection, severity of fibrosis (using non-invasive measures), and HCV detection rate in patients with End stage renal disease on hemodialysis.
2. To calculate the average treatment-lag time (time from HCV diagnosis to submission of treatment approval).

DETAILED DESCRIPTION:
This study is being conducted to evaluate real-world effectiveness of HCV DAA therapy in CHC hemodialysis patients when the DAA-treatment is managed and monitored by the nephrologist of hemodialysis center.

Hepatitis C virus (HCV) infects an estimated 185 million individuals worldwide (1) and 3.4 million to 4.4 million people in the United States.(2) Approximately 80% of acutely infected HCV patients progress to chronic infection, 20% of whom develop cirrhosis within 25 years, with 25% of patients with cirrhosis developing hepatocellular carcinoma and/or decompensated liver disease.(3) Hepatitis C virus is the primary cause of liver transplantation in the United States.(4) There are 6 known genotypes of HCV. The most common genotypes in the United States are genotype 1 (subtypes 1a and 1b), 2, and 3, which together comprise 97% of all infections.(5) Since the discovery of HCV in 1989 (6) strategies to cure the infection have evolved dramatically. A cure is defined as a sustained virologic response (SVR) and consists of undetectable levels of plasma HCV RNA 12 or 24 weeks after therapy completion.(7) Treatment of HCV has evolved rapidly and has led to improved rates of SVR.

Although these highly effective therapies for hepatitis C virus (HCV) infection have revolutionized treatment, only a few patients are able to receive treatment.(8) Barriers arising at multiple levels, from diagnosis to specialist referral, that still need to be overcome to move toward disease eradication.(9) In chronic kidney disease (CKD) patients, the prevalence of HCV infection is higher than in the general population. Testing for HCV in hemodialysis patients should be repeated every 6 months.(10) The national study on dialysis-associated diseases was published in 2002 and represents the infection statistics from dialysis center nationwide.(11) The overall estimated prevalence of HCV antibody in this study was 7.8%.

In addition, patients with impaired kidney function have limited therapeutic options. The US Food and Drug Administration (FDA) recently approved Elbasvir/Grazopevir for treatment of genotype 1 and 4 infection in CKD patients including those on hemodialysis.

At our institution, the Multidisciplinary Approach to the Treatment of Chronic Hepatitis C (MATCH) Initiative is a program which was first implemented to increase screening, diagnosis and treatment of HCV by actively incorporating primary care providers (PCP) at every step of the HCV care process. Following implementation of MATCH, early data indicates, marked increase in screening high risk and baby-boomer cohorts, as well as safe and effective treatment of HCV cases at the primary provider setting. The initiative proved that active participation of PCPs in the care of HCV reduced the treatment lag by 71% compared to traditional care of referring HCV cases to specialized care (Gastroenterology or Hepatology) while keeping similar SVR. (13) We intend to expand the program to improve quality of care for HCV patients in dialysis center. We propose active involvement of dialysis clinical staff including nephrologist, to increase HCV screening rate, promote timely diagnosis and treatment of CHC in patient with end-stage renal disease.

Rationale of the study- We will perform a phase IV study to prove real world effectiveness of Zepatier in successful treatment of CHC in patients on chronic hemodialysis at hemodialysis centers, when administered under the supervision of a nephrologist. The study will be conducted in the selected collaborative hemodialysis centers.

Zepatier Open-label Zepatier (grazoprevir 100 mg and elbasvir 50 mg) will be administered in this study.(14, 15) Zepatier is a fixed-dose combination tablet without ribavirin. GZR is an HCV NS3/4a inhibitor while EBR is an HCV NS5A inhibitor. Both grazoprevir and elbasvir are direct-acting antivirals, which together form an effective therapy for HCV and reduce the likelihood and effects of long-term liver-related HCV complications.

Zepatier has been evaluated globally in multiple phase I, II, and III trials to treat HCV. (14, 15) Randomized, placebo-controlled trials have been carried out, which led to FDA approval for Zepatier as a treatment for genotype 1 and 4 HCV.

As of July 1, 2015, a diverse population of over 1000 HCV patients has been exposed to Zepatier either as a single agent or in combination with ribavirin or sofosbuvir in phase I/II/III studies. Zepatier has been generally well tolerated at doses of 50-100 mg GZR and 50 mg EBR orally once daily. It has been comparably effective across all subgroups it has been tested in, including non-cirrhotic and/or treatment-naïve subjects. (14, 15) Headaches, fatigue, and nausea represent the most common adverse drug reactions with Zepatier.3,4 Other drug-related adverse events have included arthralgia, insomnia, diarrhea, dizziness, pyrexia, and asthenia. (14, 15) Drug-related serious adverse events are uncommon, but include allergic reactions, possible adverse interactions with other medications, or elevated liver enzymes. In past Zepatier trials, the majority of the adverse events were reversible. These adverse events are usually mild or moderate events.

The dosage in our study (100/50 mg daily) is a commonly attainable dose in clinical practice. Zepatier has shown to be safe for subjects with chronic kidney disease or who are on hemodialysis. Less than 1% of Zepatier is excreted renally. In Merck's C-SURFER, a phase 1 randomized, controlled Zepatier trial, subjects with advanced kidney disease tolerated the drug well for the required 12 weeks without dose adjustments. (16) Zepatier trials have demonstrated a 94-100% success rate achieving HCV RNA levels of <15 IU/ml after 12 weeks of treatment (SVR-12) among genotype 1 HCV patients. (14, 15) This is a prospective cohort phase IV study using multidisciplinary approach for the treatment of hepatitis C in hemodialysis patients. Hemodialysis centers will be used to deliver all HCV related care.

The study will be conducted in the selected collaborative hemodialysis centers in Philadelphia. In addition to the standard of care (SOC), all subjects with CHC will be evaluated for HCV DAA therapy: review of clinical records, assessment of the degree of liver fibrosis using FibroScan, baseline HCV virological tests, HIV and HBV screening, etc. Baseline and follow-up laboratory tests and FibroScan imaging will be performed at the Einstein lab or an alternative laboratory if requested by the patient. Baseline clinical evaluation and follow up focused H/P will be done by the nephrologist at the dialysis unit.. The study coordinator is a MATCH-D navigator and is responsible for compiling supporting documents for HCV DAA treatment request and fax it to a designated fax number (to mimic faxing to the payers in real world scenario). Local specialty pharmacy pharmacist (also a part of the MATCH-D group) will be responsible for providing hepatitis C treatment education to approved patients, ensure delivery of DAA therapy and monitoring for any drug related adverse events.

MATCH-D group will comprise of a study coordinator, study investigators, nephrologist, specialty pharmacy pharmacist, and dialysis unit . The group will meet weekly to review cases and provide recommendations on diagnosis, DAA selection and assist with HCV treatment This study will be divided to 3 phases.

1. Training study team, dialysis center clinical staff (Quarterly refresher)
2. Identifying hepatitis C patient and evaluation for treatment
3. Treatment and follow up Phase 1: Training study team and dialysis center clinical staff education All collaborative hemodialysis centers coordinator and the study team will be educated for HCV screening, work-up, treatment and study protocol in the first month of study. There will be refresher course every 3 months.

Phase 2: Identifying hepatitis C patient and evaluation for treatment

1. Patient Screening a. Every dialysis patient will be offered HCV screening every 6 months as standard of care.

   b. HCV Ab with reflex HCV viral load will be ordered.
2. Patient Identification

   1. Patients will be assessed for positive HCV Ab and detectable viral load.
   2. Nephrologist will notifythe patient with the results.
   3. Nephrologist will have the patient complete and sign HIPAA form.
   4. Nephrologist will email patient information to the study coordinator.
   5. Study coordinator is expected to keep composite record (including the above results) of all identified patients until enrollment. This record will be utilized at the Multidisciplinary Meeting.
   6. Informed consent will be obtained by the study coordinator.
   7. Basic demographic information will be collected.
3. Patient evaluation for treatment

   1. Complete blood work and FibroScan imaging will be conducted at Einstein lab or an alternative laboratory if requested by the patient.
   2. Study coordinator is expected to ensure patients have all testing completed.
   3. Study coordinator will ensure all patients are tested for FibroScan imaging using the portable FibroScan® 530 Compact system. .

This trial will enroll approximately 71 compensated cirrhotic and non-cirrhotic, Genotype 1 and 4, HCV patients who are currently on hemodialysis. Non-invasive test will be used to determine the presence or absence of cirrhosis. All excluded CHC patients will receive standard of care. Patients who have decompensated cirrhosis or hepatoma will be referred to the hepatology clinic and receive care by the hepatologist.

Study visits There will be 4 study visits in our study. Subjects may be asked to come early before dialysis session to have physical examination or Fibroscan.

Screening and Informed consent

During screening period, the following procedures and activities will be performed at hemodialysis center after the informed consent is signed:

* Review medical history and physical examination
* Review medication list
* Review laboratory data Baseline study • First laboratory tests will be performed at the Einstein lab or an alternative laboratory if requested by the patientand include: • CBC, CMP, PT/INR • HCV PCR Viral load

  * HCV PCR genotype
  * HCV NS5A RAV testing
  * HBV screening: HBsAg, HBcAb
  * HIV 1 / 2 Ab screening
  * FibroScan
  * Women of childbearing potential will have a pregnancy test at screening visit. Phase 3: Treatment and follow up 1. Treatment a. MATCH-D group will review and discuss identified CHC patients and determine those appropriate for DAA therapy through the dialysis center, and those who require referral to Liver Center based on work-up (e.g. decompensated cirrhosis).

    i. Patients appropriate for dialysis center treatment and agreeable to treatment will be enrolled in study.

    b. Meeting to occur weekly c. Study coordinator will notify the nephrologist, who saw patient, by email of the meeting decision. Subsequently, the nephrologist should notify patient of the decision and a) refer to hepatology if needed or b) explain need for treatment.

    d. Prescription along with pertinent information (e.g. lab results, fibrosis stage, etc.) will be compiled and sent to local specialty pharmacy by the study coordinator for all enrolled patients.

    e. Specialty pharmacy will:
    1. Provide education to patients about prescribed treatment.
    2. Identify potential drug interactions and notify team.
    3. Oversee delivery of medications. Provide refill reminders to patients or dialysis center staff.
    4. Monitor medication adherence.
    5. Keep "database" that is accessible to study coordinator and MATCH-D study group Specialty pharmacy will be the investigational pharmacy who is expertised in HCV care.

Initiation treatment with Zepatier All subjects will be provided with a 28-day supply of the study drug and instructed to begin treatment once all tests are done. The study coordinator will call the patient to ensure treatment has begun for HCV with Zepatier.

As with any scientific protocol, safety will be considered before treating the patients. The MATCH-D team will evaluate the patient's overall condition and make a judgment on whether initiating treatment is safe.

Zepatier for 12 weeks or 16 weeks ± Ribavirin will be used to treat HCV genotype 1, 4 in our patients and will be supplied by Merck & Co.Inc.

Statistical Methods The data will be collected using an Excel spreadsheet and analyzed with Stata 14.0 (Statacorp., College Town, TX). Descriptive statistics will be used to summarize the demographic characteristics. Screening rates, treatment rates, and treatment lag (time from detection to treatment submission) will be calculated. Categorical variables will be compared using chi square or fischer's exact test whereas continuous variables will be compared using student's t-test. SVR rates will also be compared with historical controls. P value of less than 0.05 will be considered statistically significant.

Power/Sample Size:

Power of 0.8 with a p-value of 0.05 were used a priori for sample size calculation. As was shown in C-SURFER trial recently, SVR of 99% was attained in chronic kidney disease patients including those on dialysis. Accepting a non-inferiority margin of 5% and similar expected SVR in our cohort, the sample size was calculated to be 71 patients.

Potential Benefits The subjects will get clinical benefits as the HCV treatment can prevent cirrhosis and hepatocellular carcinoma in the future. This study also has a potential to speed up treatment evaluation and the subjects may get the treatment faster.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older on day of signing the informed consent form.
* Be on long term hemodialysis at any of the selected 4 collaborative hemodialysis centers
* Have positive anti-HCV antibody titers and detectable HCV RNA level before or after the initiation of MATCH-D.
* HCV genotype 1 and 4
* Have an HCV treatment status that is one of the following:

  1. Treatment naïve: Naive to all anti-HCV treatment
  2. Prior IFN or PEG-IFN + Ribavirin Treatment failures: Null responders, Partial responders, Relapsers
  3. P/R Intolerant: Subjects were intolerant to a prior IFN or PEG-IFN

     * Ribavirin regimen, Subjects discontinued treatment prematurely and were therefore unable to complete a full course of therapy because of drug-related toxicity.

Exclusion Criteria:

* Has evidence of decompensated chronic liver disease such as presence of or history of - ascites, gastric or variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver disease
* Have Child-Pugh B or C cirrhosis (these patients will need to be referred to a hepatologist for HCV therapy)
* Have a likelihood of receiving a renal transplant or liver transplant during the study treatment period.
* Have hepatocellular carcinoma
* Have other liver disease (which require HCV therapy to be delivered under the supervision of a hepatologist)
* A patient with a life expectancy less than 12 months
* Current untreated chronic hepatitis B infection HBsAg+ patients are excluded. Note: Patients with HBcAb+ will not be excluded, but will have HBV DNA levels checked and will be monitored while on DAA therapy and medically managed as considered appropriate by the PI.
* Have HIV and currently not under Antiretroviral Therapy (ART)
* Pregnant or nursing (lactating) women
* Albumin below 3g/dL
* Platelet count below 75,000
* Unable to comply with research study visits
* Poor venous access not allowing screening laboratory collection
* Have any condition that the investigator considers a contraindication to study participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
HCV treatment-lag time | 12 weeks
  To determine the average treatment-lag time (time from HCV diagnosis to submission of treatment approval) of HCV treatment delivered through hemodialysis centers by nephrologists compared to standard of care via traditional gastroenterology or hepatology centers.

SECONDARY OUTCOMES:
Prevalence rates | 12 weeks
  To estimate prevalence of HCV infection, severity of fibrosis (using non-invasive measures), and HCV detection rate in patients with End stage renal disease on hemodialysis.
Sustained virologic response (SVR) rates | 6 months
  2. To determine sustained virologic response (SVR) rates of open-label Zepatier in chronic hepatitis C infected (CHC) patient who are currently on hemodialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Eyob Feyssa, MD, Principal Investigator — Albert Einstein Healthcare Network; Eyob Feyssa, MD, Study Chair — Albert Einstein Healthcare Network

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shepard CW, Finelli L, Alter MJ. Global epidemiology of hepatitis C virus infection. Lancet Infect Dis. 2005 Sep;5(9):558-67. doi: 10.1016/S1473-3099(05)70216-4. PMID 16122679
- [Background] Chak E, Talal AH, Sherman KE, Schiff ER, Saab S. Hepatitis C virus infection in USA: an estimate of true prevalence. Liver Int. 2011 Sep;31(8):1090-101. doi: 10.1111/j.1478-3231.2011.02494.x. Epub 2011 Mar 16. PMID 21745274
- [Background] Freeman AJ, Dore GJ, Law MG, Thorpe M, Von Overbeck J, Lloyd AR, Marinos G, Kaldor JM. Estimating progression to cirrhosis in chronic hepatitis C virus infection. Hepatology. 2001 Oct;34(4 Pt 1):809-16. doi: 10.1053/jhep.2001.27831. PMID 11584380
- [Background] Davis GL, Alter MJ, El-Serag H, Poynard T, Jennings LW. Aging of hepatitis C virus (HCV)-infected persons in the United States: a multiple cohort model of HCV prevalence and disease progression. Gastroenterology. 2010 Feb;138(2):513-21, 521.e1-6. doi: 10.1053/j.gastro.2009.09.067. Epub 2009 Oct 25. PMID 19861128
- [Background] Delwart E, Slikas E, Stramer SL, Kamel H, Kessler D, Krysztof D, Tobler LH, Carrick DM, Steele W, Todd D, Wright DJ, Kleinman SH, Busch MP; NHLBI-REDS-II Study Group. Genetic diversity of recently acquired and prevalent HIV, hepatitis B virus, and hepatitis C virus infections in US blood donors. J Infect Dis. 2012 Mar 15;205(6):875-85. doi: 10.1093/infdis/jir862. Epub 2012 Jan 31. PMID 22293432
- [Background] Choo QL, Kuo G, Weiner AJ, Overby LR, Bradley DW, Houghton M. Isolation of a cDNA clone derived from a blood-borne non-A, non-B viral hepatitis genome. Science. 1989 Apr 21;244(4902):359-62. doi: 10.1126/science.2523562.
- [Background] Swain MG, Lai MY, Shiffman ML, Cooksley WG, Zeuzem S, Dieterich DT, Abergel A, Pessoa MG, Lin A, Tietz A, Connell EV, Diago M. A sustained virologic response is durable in patients with chronic hepatitis C treated with peginterferon alfa-2a and ribavirin. Gastroenterology. 2010 Nov;139(5):1593-601. doi: 10.1053/j.gastro.2010.07.009. Epub 2010 Jul 14. PMID 20637202
- [Background] McGowan CE, Fried MW. Barriers to hepatitis C treatment. Liver Int. 2012 Feb;32 Suppl 1(0 1):151-6. doi: 10.1111/j.1478-3231.2011.02706.x. PMID 22212587
- [Background] Konerman MA, Lok AS. Hepatitis C Treatment and Barriers to Eradication. Clin Transl Gastroenterol. 2016 Sep 22;7(9):e193. doi: 10.1038/ctg.2016.50. PMID 27657495
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO). KDIGO clinical practice guidelines for the prevention, diagnosis, evaluation, and treatment of hepatitis C in chronic kidney disease. Kidney Int Suppl. 2008 Apr;(109):S1-99. doi: 10.1038/ki.2008.81. No abstract available. PMID 18382440
- [Background] Finelli L, Miller JT, Tokars JI, Alter MJ, Arduino MJ. National surveillance of dialysis-associated diseases in the United States, 2002. Semin Dial. 2005 Jan-Feb;18(1):52-61. doi: 10.1111/j.1525-139X.2005.18108.x. PMID 15663766
- [Background] AASLD/IDSA HCV Guidance Panel. Hepatitis C guidance: AASLD-IDSA recommendations for testing, managing, and treating adults infected with hepatitis C virus. Hepatology. 2015 Sep;62(3):932-54. doi: 10.1002/hep.27950. Epub 2015 Aug 4. No abstract available. PMID 26111063
- [Background] Sandhu N, Mulki R, Tosounian S, Wheeler D, Feyssa E, Baumann A. Multidisciplinary Approach to the Treatment of Chronic Hepatitis C: The MATCH Initiative AASLD Abstract presentation. 2017.
- [Background] Forns X, Gordon SC, Zuckerman E, Lawitz E, Calleja JL, Hofer H, Gilbert C, Palcza J, Howe AY, DiNubile MJ, Robertson MN, Wahl J, Barr E, Buti M. Grazoprevir and elbasvir plus ribavirin for chronic HCV genotype-1 infection after failure of combination therapy containing a direct-acting antiviral agent. J Hepatol. 2015 Sep;63(3):564-72. doi: 10.1016/j.jhep.2015.04.009. Epub 2015 Apr 18. PMID 25895428
- [Background] Zeuzem S, Ghalib R, Reddy KR, Pockros PJ, Ben Ari Z, Zhao Y, Brown DD, Wan S, DiNubile MJ, Nguyen BY, Robertson MN, Wahl J, Barr E, Butterton JR. Grazoprevir-Elbasvir Combination Therapy for Treatment-Naive Cirrhotic and Noncirrhotic Patients With Chronic Hepatitis C Virus Genotype 1, 4, or 6 Infection: A Randomized Trial. Ann Intern Med. 2015 Jul 7;163(1):1-13. doi: 10.7326/M15-0785. PMID 25909356
- [Background] Roth D, Nelson DR, Bruchfeld A, Liapakis A, Silva M, Monsour H Jr, Martin P, Pol S, Londono MC, Hassanein T, Zamor PJ, Zuckerman E, Wan S, Jackson B, Nguyen BY, Robertson M, Barr E, Wahl J, Greaves W. Grazoprevir plus elbasvir in treatment-naive and treatment-experienced patients with hepatitis C virus genotype 1 infection and stage 4-5 chronic kidney disease (the C-SURFER study): a combination phase 3 study. Lancet. 2015 Oct 17;386(10003):1537-45. doi: 10.1016/S0140-6736(15)00349-9. Epub 2015 Oct 5. PMID 26456905
- [Background] Merck Sharp & Dohme Corporation (January 2016). ZEPATIER™ tablets. Highlights of Prescribing Information. 2016.
- [Background] Merck Sharp & Dohme Corporation (July 2015). Elbasvir (MK-8742). Investigator's Brochure (8th Ed.).2015.
- [Background] Merck Sharp & Dohme Corporation (July 2015). Grazoprevir (MK-5172). Investigator's Brochure (10th Ed.). 2015.